CLINICAL TRIAL: NCT03065920
Title: African Severe Asthma Program
Brief Title: African Severe Asthma Program: A Research Network for Characterisation of Severe Asthma in Africans (ASAP)
Acronym: ASAP
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, Bruce J Kirenga, Dr Bruce J Kirenga, Makerere University
Other Study IDs: ASAP 001
Record Dates: First submitted 2016-08-18; First posted 2017-02-28 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Replicative single nucleotide polymorphisms (SNP) genotying: Subjects enrolled into the study will be invited to participate in genetic research by providing a blood sample.
  DNA will be extracted from the blood samples.Part of the DNA will be used for replicative severe asthma associated SNPs genotying of SNPs previously reported to be associated with severe asthma. The remaining samples will be biobanked for future genetic and pharmacogenetic studies.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a prospective observational multicentre cohort study of asthma patients in Eastern Africa whose objectives will be; The primary objective of this project is to identify and characterize severe asthma in Eastern Africa in order to understand its demographic, clinical, physiologic, pathologic, genomic and immunologic determinants.

Secondary objective(s) are; Compare the annual healthcare utilisation (HCU) (emergency room visits, hospitalization including admission to critical care units and unscheduled outpatient clinic or office visits), exacerbation, quality of life and mortality rates of severe and not- severe asthma patients Determine the factors associated with the asthma HCU events, quality of life, exacerbations and mortality The study will enroll 1676 patients aged between 12 and 70 years and follow up each patient for up to one year.

DETAILED DESCRIPTION:
This study is a prospective observational multicentre cohort study of asthma patients in Eastern Africa. whose objectives will be; The primary objective of this project is to identify and characterize severe asthma in Eastern Africa in order to understand its demographic, clinical, physiologic, pathologic, genomic and immunologic determinants.

Secondary objective(s) are; Compare the annual healthcare utilisation (HCU) (emergency room visits, hospitalization including admission to critical care units and unscheduled outpatient clinic or office visits), exacerbation, quality of life and mortality rates of severe and not- severe asthma patients Determine the factors associated with the asthma HCU events, quality of life, exacerbations and mortality.

The study will enroll 1676 patients aged between 12 and 70 years and follow up each patient for up to one year.

Measurements; The following will be done

* Asthma Diagnosis. This will be done and will be an entry point to the study. It will be done to ensure patients enrolled onto the study fulfill a clinical diagnosis of Asthma.
* Cohort Characterisation. Through use of a predeveloped clinical review form, data on demographics, symptoms, exposures to pollutants, known asthma triggers, tobacco smoking, psychosocial issues, comorbidities, asthma control, adherence to medication and inhaler technique will be collected. Asthma quality of life will also be ascertained through use of a questionnaire.

Further measurements to characterise asthma will be performed and include;

* Spirometry
* Bronchial hyperresponsiveness testing using methacholine challenge tests
* Skin prick test (SPT), total IgE assays and complete blood count (for eosinophils)
* FeNO for airway inflammation according to published guidelines.
* Stool microscopy for helminths infestation
* Replicative single nucleotide polymorphisms (SNP) genotying
* HIV testing Each patient will be followed up at intervals (initially monthly for 6 months and then at month 9 and 12). At each clinic visit, treatment will be optimised.

ELIGIBILITY:
Inclusion Criteria:

* All Asthma Patients presenting at study clinics who are between 12 and 70 years and older resident within 30km of the enrolling sites.

Exclusion Criteria:

* Asthma patients with contra-indications to any of the study procedures and tests.

In addition the following patients will be excluded:

* Patients with a primary diagnosis of an alternative lung disease (e.g.: COPD, or bronchiectasis, pulmonary fibrosis.),
* Patients with another significant disease likely to confound assessment of asthma (e.g: active tuberculosis),
* Patients unable to perform study tests and procedures,
* Patients over 70 years of age, patients who have been exposed to experimental treatments within the past three months
* Pregnant women.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All Asthma Patients presenting at study clinics during the study period. These will have to be 12 years and older resident within 30km radius 'of the enrolling sites.
  Asthma will be defined as either doctor diagnosed, clinical/treated asthma and wheezing/whistling breath in the last 12 months as used in the World Health Survey and other surveys.
Sampling Method: Non-Probability Sample
Enrollment: 1676 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with Severe Asthma. | 3 years
  The primary end point in this study is severe asthma. We shall document the proportion of the enrolled patients that have severe asthma and perform a factor analysis to identify factors independently associated with severe asthma.

SECONDARY OUTCOMES:
Treatment Severe Asthma | 3 years
  Incidences rates of this outcome between groups (severe and not severe asthma) will be compared and predictors of this outcome analysed.
Health Care Utilisation rates | 3 years
  Incidences rates of this outcome between groups (severe and not severe asthma) will be compared and predictors of this outcome analysed.
Exacerbations | 3 years
  Incidences rates of this outcome between groups (severe and not severe asthma) will be compared and predictors of this outcome analysed.
Mortality rates | 3 years
  Incidences rates of this outcome between groups (severe and not severe asthma) will be compared and predictors of this outcome analysed.

CONTACTS AND LOCATIONS:
Locations (4):
- Black Lion Hospital, Addis Ababa, Central, Ethiopia
- Kenyatta National Hospital, Nairobi, Central, Kenya
- Groningen Research Institute for Asthma and COPD (GRIAC), Amsterdam, Central, Netherlands
- Mulago Hospital, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kwizera R, Bongomin F, Olum R, Worodria W, Bwanga F, Meya DB, Kirenga BJ, Gore R, Denning DW, Fowler SJ. Evaluation of an Aspergillus IgG/IgM lateral flow assay for serodiagnosis of fungal asthma in Uganda. PLoS One. 2021 May 28;16(5):e0252553. doi: 10.1371/journal.pone.0252553. eCollection 2021. PMID 34048497
- [Derived] Kwizera R, Wadda V, Mugenyi L, Aanyu-Tukamuhebwa H, Nyale G, Yimer G, Chakaya J, De Jong C, Van der Molen T, Denning DW, Gore R, Kirenga BJ. Skin prick reactivity among asthmatics in East Africa. World Allergy Organ J. 2020 Jun 23;13(6):100130. doi: 10.1016/j.waojou.2020.100130. eCollection 2020 Jun. PMID 32612738